CLINICAL TRIAL: NCT06136988
Title: A Multicenter, Open-label, Phase Ib/II Study of Docetaxel for Injection (Albumin-bound) and SG001 in Combination With Cisplatin and Simultaneous Radiotherapy Versus Paclitaxel in Combination With Cisplatin and Simultaneous Radiotherapy for Locally Advanced Unresectable Esophageal Squamous Carcinoma.
Brief Title: A Study of Docetaxel for Injection (Albumin-bound) and SG001 in Combination With Cisplatin and Simultaneous Radiotherapy for Locally Advanced Unresectable Esophageal Squamous Carcinoma.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB1801-008
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Locally Advanced Unresectable Esophageal Squamous Carcinoma
MeSH Terms: interventions — Docetaxel; Injections; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HB1801 and SG001 in combination with cisplatin and simultaneous radiotherapy (Experimental): SG001 360 mg, Intravenous infusion, D1, Q3W, up to approximately 2 years ; Docetaxel for Injection (Albumin-bound) (HB1801), Intravenous infusion, D1, Q3W, 60 or 75 mg/m^2, up to 2 cycles; cisplatin for injection 25 mg/m^2, D1-D3, Q3W, up to 2 cycles; radiotherapy (28×1.8Gy).All treatments will be administered until disease progression or intolerable toxicity.
  Interventions: Drug: Docetaxel for Injection (Albumin-bound); Drug: SG001; Drug: Cisplatin for injection; Radiation: Simultaneous Radiotherapy
- Paclitaxel in combination with cisplatin and simultaneous radiotherapy (Active Comparator): Paclitaxel 135 mg/m^2, Intravenous infusion, D1, Q3W; cisplatin for injection 25 mg/m^2, D1-D3, Q3W, radiotherapy (28×1.8Gy). No other systemic antineoplastic therapy is allowed until disease progression, optimal supportive care and local palliative care are allowed.
  Interventions: Drug: Cisplatin for injection; Drug: Paclitaxel; Radiation: Simultaneous Radiotherapy

INTERVENTIONS:
Drug: Docetaxel for Injection (Albumin-bound) — Docetaxel for Injection (Albumin-bound) 60 or 75 mg/m^2, Intravenous infusion, Q3W
  Other Names: HB1801
  Arms: HB1801 and SG001 in combination with cisplatin and simultaneous radiotherapy
Drug: SG001 — Recombinant Anti-PD-1 Fully Human Monoclonal Antibody Injection, 360 mg, Intravenous infusion, Q3W
  Other Names: Recombinant Anti-PD-1 Fully Human Monoclonal Antibody Injection
  Arms: HB1801 and SG001 in combination with cisplatin and simultaneous radiotherapy
Drug: Cisplatin for injection — Cisplatin for injection, 25 mg/m^2, Intravenous infusion, D1-D3, Q3W
Drug: Paclitaxel — Paclitaxel 135 mg/m^2, Intravenous infusion, Q3W
  Arms: Paclitaxel in combination with cisplatin and simultaneous radiotherapy
Radiation: Simultaneous Radiotherapy — Radiotherapy (28×1.8Gy)

SUMMARY:
The study is a multicenter, open-label, phase Ib/II study to evaluate the efficacy and safety of docetaxel for injection (albumin-bound) (HB1801) and SG001 in combination with cisplatin and simultaneous radiotherapy versus paclitaxel in combination with cisplatin and simultaneous radiotherapy for locally advanced unresectable esophageal squamous carcinoma.

DETAILED DESCRIPTION:
This study will be conducted in two stages. The first stage (Phase Ib) is a dose-escalation study designed to determine the safety and the recommended Phase 2 dose (RP2D) of HB1801 and SG001 in combination with cisplatin and simultaneous radiotherapy for locally advanced unresectable esophageal squamous carcinoma. Patients will be assigned to receive sequentially higher doses of HB1801 once every three weeks (a Cycle) by intravenous infusion, starting at a dose of 60 mg/m^2. The second stage (Phase II) is a study to evaluate the efficacy and safety of HB1801 and SG001 in combination with cisplatin and simultaneous radiotherapy versus paclitaxel in combination with cisplatin and simultaneous radiotherapy for locally advanced unresectable esophageal squamous carcinoma. Regular visits and imaging examinations will be conducted to compare the efficacy and safety of the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years (based on the day of signing the informed consent form).
2. Voluntarily sign the informed consent, willing and able to follow the protocol for visits, treatment and laboratory tests.
3. Locally advanced (stage II-IVa and IVb supraclavicular lymph node metastases according to AJCC 8th edition) esophageal squamous carcinoma (in the case of mixed adenosquamous carcinoma, more than 50% squamous carcinoma component can be screened) diagnosed histologically or cytologically, which is unresectable in the judgment of the principal investigator, and is amenable to definitive chemoradiotherapy (dCRT) .
4. ECOG score of 0-1 within 7 days prior to the first dose.
5. Vital organ function within 7 days prior to first dose, meeting the following criteria (no blood transfusions, no use of human granulocyte colony-stimulating factor (G-CSF), thrombopoietin (TPO), and erythropoietin (EPO) within 14 days prior to the first dose):

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   2. Platelet count (PLT) ≥ 100×10^9/L
   3. Hemoglobin ≥ 80g/L
   4. Serum albumin ≥ 28g/L
   5. Total bilirubin ≤1.0×ULN; ALT/AST ≤1.5×ULN
   6. Serum creatinine ≤1.5×ULN or creatinine clearance ≥60 mL/min, Cockcroft-Gault formula
   7. Activated Prothrombin Time (APTT) and International Normalized Ratio (INR) ≤ 1.5 x ULN.
6. Female patients of childbearing age tested negative serum pregnancy test within 7 days prior to the first dose, and patients must agree to take effective contraception from the signing of the informed consent form until 6 months after the last dose, during which time breastfeeding is not allowed; male patients must agree to take contraception and sperm donation is not allowed.
7. Have at least one evaluable lesion per Response Evaluation Criteria In Solid Tumors (RECIST 1.1).

Exclusion Criteria:

1. Active malignancy within 5 years prior to the first dose, except esophageal carcinoma studied in this trial and any locally curable tumor that has received radical therapy (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or early-stage thyroid cancer, etc).
2. History of esophageal perforation and/or esophageal fistula within 6 months prior to the first dose; or significant tumor invasion into an organ adjacent to the esophageal lesion (aorta or trachea), etc., resulting in a high risk of hemorrhage, esophageal fistula, or signs of esophageal perforation.
3. Uncontrollable plasma effusions requiring frequent drainage or medical intervention (e.g., pleural effusion, peritoneal effusion, pericardial effusion, etc.) within 7 days prior to the first dose that require additional interventions within 2 weeks of the intervention (excluding exfoliative cytology of the exudate).
4. Weight loss of 20% or more within 3 months prior to the first dose; or BMI <18.5 kg/m^2 and/or weight <30 kg.
5. Severe allergy history to albumin or docetaxel, paclitaxel, cisplatin, or monoclonal antibody drugs.
6. Patients who have received prior antitumor therapy for esophageal cancer.
7. Patients with immunodeficiency or active autoimmune disease (except a. well-controlled type I diabetes b. hypothyroidism [controlled with hormone replacement therapy] c. well-controlled celiac disease d. dermatologic that do not require systemic therapy [e.g., vitiligo, psoriasis, alopecia] e. any other condition not expected to recur in the absence of external triggers).
8. History of severe cardiovascular disease within 6 months prior to the first dose, including but not limited to:

   1. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, Third-degree atrioventricular block
   2. History of myocardial infarction, unstable angina, angioplasty, coronary artery bridging surgery
   3. Heart failure with New York Heart Association (NYHA) classification of class III and above
   4. Left ventricular ejection fraction (LVEF) <50% at screening period
   5. Patients with prolonged QT/QTc interval on ECG at baseline (QTcF > 480ms, Fridericia formula: QTcF=QT/RR^0.33, RR=60/heart rate).
9. Patients with poorly controlled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg during the screening period).
10. Patients with active Hepatitis B (Hepatitis B surface antigen (HBsAg) or HBcAb positive test and active stage of Hepatitis B (HBV-DNA ≥ 10^4 cps/mL or ≥ 2000 IU/mL)); Hepatitis C (Hepatitis C Antibody (Anti-HCV) positive test and a positive PCR result for HCV RNA); positive for HIV, during the screening period.
11. Patients with poorly controlled diabetes mellitus, or hypokalemia, hyponatremia, or abnormal values on corrected calcium lab tests (CTCAE 5.0 >1 grade) despite of standard drug therapy within 14 days prior to the first dose.
12. History of interstitial lung disease or non-infectious pneumonia.
13. Patients with known psychoneurologic disorders that may affect adherence to the trial, and those with a history of drug dependence;
14. Patients with severe chronic or active infections (including tuberculosis infection, etc.) requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days prior to the first dose. Note: Antiviral therapy for patients with viral hepatitis is permitted.
15. Have received potent inhibitors or potent inducers of CYP2C8 (for Phase Ⅱ trials only) or CYP3A4 within 14 days prior to the first dose.
16. Vaccination with a live or live attenuated vaccine (inactivated vaccines are permitted) within 28 days prior to the first dose.
17. History of major organ surgery (excluding puncture biopsy) within 28 days prior to the first dose.
18. Patients who have received antitumor therapy such as other clinical investigational drugs within 28 days prior to the first dose.
19. Patients who have received systemic glucocorticoid therapy (dose > 10 mg/day of prednisone or equivalent) within 28 days prior to the first dose.
20. Any condition that, in the opinion of the investigator, makes participation in the study inappropriate (including, but not limited to, concurrent serious or uncontrolled medical conditions, potential safety risks, interference with the interpretation of the results of the study, and adherence to the trial).
21. The patient is concurrently participating in another clinical study, unless it is an observational (non-interventional) clinical study or is in the follow-up period of an interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 21 days)
Determine the recommended Phase 2 dose (RP2D) of Docetaxel for Injection (Albumin-bound) | At the end of Cycle 2 (each cycle is 21 days)
Incidence and frequency of adverse events (AE) and serious adverse events (SAE) in Phase Ib | up to 4 years
PFS as determined by the investigator according to RECIST 1.1 in Phase Ⅱ | up to 4 years

SECONDARY OUTCOMES:
Objective remission rate (ORR) | up to 4 years
Disease control rate (DCR) | up to 4 years
Duration of remission (DOR) | up to 4 years
Progression-free survival (PFS) | up to 4 years
Overall survival (OS) | up to 4 years
Incidence of SG001 antidrug antibodies and neutralizing antibodies (if applicable) | up to 4 years
Incidence and frequency of adverse events (AE) and serious adverse events (SAE) in Phase Ⅱ | up to 4 years

OTHER OUTCOMES:
Total docetaxel concentration in plasma and free docetaxel concentration | up to 4 years
SG001 concentration in serum | up to 4 years
To evaluate the correlation between PD-L1 expression and efficacy in tumor tissues | up to 4 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shandong Tumor Hospital, Jinan, Shandong
  - Tianjin cancer institute &hospital, Tianjin, Tianjin Municipality